CLINICAL TRIAL: NCT01012895
Title: Parallel, Open-Label, Randomized, Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-790052 and BMS-650032 in Combination in Null Responders to Standard of Care Infected With Chronic Hepatitis C Virus Genotype 1
Brief Title: Study to Determine the Effectiveness of Antiviral Combination Therapy to Treat Hepatitis C Virus (HCV) Infected Patients Who Have Previously Failed Standard of Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI447-011; 2010-024637-23 (EudraCT Number)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir; asunaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Arm 1: Sentinel A (Experimental): BMS-790052 (60mg) once daily + BMS-650032 (600 mg) twice daily
  Interventions: Drug: BMS-790052; Drug: BMS-650032
- Arm 2: Sentinel B (Experimental): BMS-790052 (60mg) once daily + BMS-650032 (600mg) twice daily + Pegylated-interferon alfa-2a + Ribavirin
  Interventions: Drug: BMS-790052; Drug: BMS-650032; Drug: Pegylated-interferon alfa-2a; Drug: Ribavirin
- Arm 3: Expansion A1 (Experimental): BMS-790052 (60mg) once daily + BMS-650032 (200mg) twice daily
  Interventions: Drug: BMS-790052; Drug: BMS-650032
- Arm 4: Expansion A2 (Experimental): BMS-790052 (60mg) once daily + BMS-650032 (200mg) once daily
  Interventions: Drug: BMS-790052; Drug: BMS-650032
- Arm 5: Expansion B1 (Experimental): BMS-790052 (60mg) once daily + BMS-650032 (200 mg) twice daily + Pegylated-interferon alfa-2a + Ribavirin
  Interventions: Drug: BMS-790052; Drug: BMS-650032; Drug: Pegylated-interferon alfa-2a; Drug: Ribavirin
- Arm 6: Expansion B2 (Experimental): BMS-790052 (60mg) once daily + BMS-650032 (200 mg) once daily + Pegylated-interferon alfa-2a + Ribavirin
  Interventions: Drug: BMS-790052; Drug: BMS-650032; Drug: Pegylated-interferon alfa-2a; Drug: Ribavirin
- Arm 7: Expansion B3 (Experimental): BMS-790052 (60 mg) once daily + BMS-650032 (200 mg) twice daily + Ribavirin
  Interventions: Drug: BMS-790052; Drug: BMS-650032; Drug: Ribavirin

INTERVENTIONS:
Drug: BMS-790052 — Tablets, Oral, 60 mg, once daily, 24 weeks
Drug: BMS-650032 — Tablets, Oral, 600 mg, twice daily, 24 weeks
  Arms: Arm 1: Sentinel A; Arm 2: Sentinel B
Drug: BMS-650032 — Tablets, Oral, 200mg, twice daily, 24 weeks
  Arms: Arm 3: Expansion A1; Arm 5: Expansion B1; Arm 7: Expansion B3
Drug: BMS-650032 — Tablets, Oral, 200 mg, once daily, 24 weeks
  Arms: Arm 4: Expansion A2; Arm 6: Expansion B2
Drug: Pegylated-interferon alfa-2a — Syringe, Subcutaneous Injection, 180 µg, once weekly
  Other Names: Pegasys
  Arms: Arm 2: Sentinel B; Arm 5: Expansion B1; Arm 6: Expansion B2
Drug: Ribavirin — Tablets, Oral
  For subjects weighing < 75 kg: 1000 mg; For subjects weighing ≥ 75 kg: 1200 mg
  Twice daily (< 75 kg: 400 mg in ante meridian (AM) and 600 mg in post meridian (PM); ≥ 75 kg: 600 mg in AM and PM), 24 weeks
  Other Names: Copegus
  Arms: Arm 2: Sentinel B; Arm 5: Expansion B1; Arm 6: Expansion B2; Arm 7: Expansion B3

SUMMARY:
The purpose of this study is to determine whether BMS-650032 and BMS-790052 in combination alone, together with Ribavirin, or together with Interferon and Ribavirin are effective in the treatment of Hepatitis C in patients who have not responded to prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18 to 70 years
* HCV-Infected Genotype 1 Null responders to current standard of care
* Expansion Cohorts A1 and A2 are restricted to patients infected with HCV Genotype 1b only.

Exclusion Criteria:

* Evidence of a medical condition associate with chronic liver disease other than HCV
* History of variceal bleeding, hepatic encephalopathy, or ascites requiring management with diuretics or paracentesis
* History of Cancer within 5 years of enrollment
* History of gastrointestinal disease or surgical procedure (except Cholecystectomy)
* History of clinically significant cardiac disease
* History of Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Documented cirrhosis within 12 months prior to dosing
* Positive for Human Immunodeficiency Virus (HIV) or Hepatitis B Virus (HBV)
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Hepatitis C virus (HCV) ribonucleic acid (RNA) levels in subjects' blood before, during and after treatment | 12 weeks post treatment

SECONDARY OUTCOMES:
Safety assessments will be based on medical review of the frequency of SAEs and AEs, discontinuations due to AEs, and abnormalities observed from vital sign and ECG measurements, physical examinations and clinical laboratory results | 12 weeks post-treatment
  Serious Adverse Events (SAEs), Adverse Events (AEs), Electrocardiogram (ECG)
Pharmacokinetic parameter maximum observed concentration [Cmax] will be derived from plasma concentration versus time. Trough concentration (Ctrough) and sparse Pharmacokinetics (PK) samples will also be collected. | Day 1 and Day 14
Pharmacokinetic parameter trough observed concentration [Cmin] will be derived from plasma concentration versus time. Trough concentration (Ctrough) and sparse Pharmacokinetics (PK) samples will also be collected. | Days 1, Days 7, Days 14, Weeks 4, Weeks 8, Weeks 12, Weeks 16
Pharmacokinetic parameter time of maximum observed concentration [Tmax] will be derived from plasma concentration versus time. Trough concentration (Ctrough) and sparse Pharmacokinetics (PK) samples will also be collected. | Day 1 and Day 14
Pharmacokinetic parameter area under the concentration-time curve in one dosing interval [AUC(TAU)] will be derived from plasma concentration versus time. Trough concentration (Ctrough) and sparse Pharmacokinetics (PK) samples will also be collected. | Day 1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (10):
  - Advanced Clinical Research Institute, Anaheim, California
  - Southern California Liver Centers, Coronado, California
  - San Jose Gastroenterology, San Jose, California
  - University Of Colorado Denver & Hospital, Aurora, Colorado
  - Mercy Medical Center, Baltimore, Maryland
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - Texas Clinical Research Institute, Llc, Arlington, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
- France (5):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Pessac
- Local Institution, San Juan, Puerto Rico

REFERENCES:
- [Derived] Kao JH, Jensen DM, Manns MP, Jacobson I, Kumada H, Toyota J, Heo J, Yoffe B, Sievert W, Bessone F, Peng CY, Roberts SK, Lee YJ, Bhore R, Mendez P, Hughes E, Noviello S. Daclatasvir plus asunaprevir for HCV genotype 1b infection in patients with or without compensated cirrhosis: a pooled analysis. Liver Int. 2016 Jul;36(7):954-62. doi: 10.1111/liv.13049. Epub 2016 Jan 24. PMID 26683763
- [Derived] McPhee F, Hernandez D, Yu F, Ueland J, Monikowski A, Carifa A, Falk P, Wang C, Fridell R, Eley T, Zhou N, Gardiner D. Resistance analysis of hepatitis C virus genotype 1 prior treatment null responders receiving daclatasvir and asunaprevir. Hepatology. 2013 Sep;58(3):902-11. doi: 10.1002/hep.26388. Epub 2013 Jul 16. PMID 23504694
- [Derived] Lok AS, Gardiner DF, Lawitz E, Martorell C, Everson GT, Ghalib R, Reindollar R, Rustgi V, McPhee F, Wind-Rotolo M, Persson A, Zhu K, Dimitrova DI, Eley T, Guo T, Grasela DM, Pasquinelli C. Preliminary study of two antiviral agents for hepatitis C genotype 1. N Engl J Med. 2012 Jan 19;366(3):216-24. doi: 10.1056/NEJMoa1104430. PMID 22256805
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx